CLINICAL TRIAL: NCT05302518
Title: Virtual Reality for AnxIety Disorders - Randomized Controlled Trial
Acronym: VR8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region of Southern Denmark (Other)
Collaborators: University of Southern Denmark (Other); Odense University Hospital (Other); Universite du Quebec en Outaouais (Other); IMotions A/S (Industry)
Responsible Party: Principal Investigator, Per T Ørskov, Postdoc, Region of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21/59870; 9069-00043B (Other Grant/Funding Number: Innovation Fund Denmark)
Record Dates: First submitted 2022-03-09; First posted 2022-03-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Social Anxiety; Social Phobia
Keywords: Social anxiety; Cognitive behavioral therapy; Virtual reality; Exposure; Psychophysiological Measurement; Heart Rate; Electrodermal Activity
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive behavioral therapy with exposure in virtual reality (Experimental): This arm of the study will receive cognitive behavioral therapy with exposure in virtual reality. The intervention is individual and manualized and delivered by a psychologist. The intervention consists of 10 weekly session with a duration of 60 minutes. Exposure is conducted from session 4 to 9. Homework is assigned and it includes exposure in vivo. The amount of exposure is controlled for.
  Interventions: Behavioral: Cognitive behavioral therapy with exposure in virtual reality
- Cognitive behavioral therapy with exposure in vivo (Active Comparator): This arm of the study will receive cognitive behavioral therapy with exposure in vivo. The intervention is individual and manualized and delivered by a psychologist. The intervention consists of 10 weekly session with a duration of 60 minutes. Exposure is conducted from session 4 to 9. Homework is assigned and it includes exposure in vivo. The amount of exposure is controlled for.
  Interventions: Behavioral: Cognitive behavioral therapy with exposure in vivo

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy with exposure in virtual reality — The treatment rationale is based on a model of the maintenance of social phobia by Clark and Wells. The themes of therapy are: a) The general ideas of CBT, b) The maintaining processes of social phobia, c) negative automatic thoughts, d) shifting focus of attention form self-focus to external focus, e) safety behaviors, f) post-processing, g) self-processing, h) schemas and rules for living.
  Exposure in VR:
  We will use 360° 3D videos for exposure using an HTC Vive Pro headset. Six different videos will be used for exposure: 1) Taking a seat on a bench in a public park, 2) Being introduced as a new employee, 3) Performing a presentation at a meeting, 4) Entering and shopping in a grocery store, 5) Visiting a café and 6) Using public transportation. The therapist can choose the length of the exposure as well as the difficulty of the exposure. While the participant is in the VR-scenario HR and EDA are measured. These data are collected to continuously estimate the anxiety levels.
  Other Names: CBT-ExpVR
  Arms: Cognitive behavioral therapy with exposure in virtual reality
Behavioral: Cognitive behavioral therapy with exposure in vivo — The treatment rationale is based on a model of the maintenance of social phobia by Clark and Wells.The themes of therapy are: a) The general ideas of CBT, b) The maintaining processes of social phobia, c) negative automatic thoughts, d) shifting focus of attention form self-focus to external focus, e) safety behaviors, f) post-processing, g) self-processing, h) schemas and rules for living.
  Exposure in vivo:
  Exposure is taking place at Centre for Telepsychiatry and the surrounding areas. The therapist is planning the exposure with the participant and is accompanying the participant during the exposure.
  Other Names: CBT-Exp
  Arms: Cognitive behavioral therapy with exposure in vivo

SUMMARY:
Social anxiety disorder (SAD) has a high prevalence and an early onset and has a lengthy recovery period often taking decades to occur. Current evidence supports the efficacy of cognitive behavioral therapy (CBT) with virtual reality (VR) exposure. However, the evidence is based on a small number of studies.

This trial examines the efficacy of an intervention that combines CBT with individually tailored exposure in VR. During exposure, participants' anxiety level is estimated in real time based on heart rate and electrodermal activity. Estimated anxiety level can guide the therapist's adjustment of the VR content. The above treatment is compared with the gold standard treatment for SAD which is cognitive behavioral therapy with exposure conducted in real life. Treatment is individual, manual-based and consists of 10 weekly sessions with a duration of 60 minutes.

The aim of the study is to investigate whether CBT combined with exposure in VR (adapted on the basis of estimated anxiety level) is more effective than CBT with exposure in real life.

The trial is a randomized controlled trail (RCT). The study includes 90 participants diagnosed with SAD. Assessments are carried out pre-treatment, mid-treatment and at follow-up (6 and 12 months).

The primary outcome of the study is self-reported symptoms of social anxiety using Social Interaction Anxiety Scale. The primary endpoint is post-treatment.

DETAILED DESCRIPTION:
INTRODUCTION

Social anxiety disorder (SAD) is a common anxiety disorder characterized by excessive fear of being scrutinized or criticized by others leading to avoidance of social situations. According to the ICD-10 classification of mental and behavioral disorders, engaging in feared situations is accompanied by autonomic symptoms of anxiety such as sweating, trembling or increased heartrate (HR). The lifetime prevalence of SAD ranges between 8.4% and 12.1% and the 12 month prevalence ranges between 4.2% and 7.1%.

SAD is related to reduced health-related quality of life and is also associated with substantial psychiatric comorbidity including other anxiety disorders, mood disorders and substance use disorders. Epidemiological studies show that SAD most often precedes depression and that SAD is related to a substantially and consistently increase in risk of subsequent depression. Similarly, symptoms of social anxiety often precedes alcohol dependence.

SAD is an adolescent-onset disorder with a long recovery period. Despite the prolonged recovery, few individuals with SAD seek treatment for their disorder. Only about one-third of lifetime cases report ever seeking treatment for SAD. Not seeking treatment may be related to the nature of the disorder itself. Individuals with SAD avoid treatment because the treatment itself constitutes a social situation that provokes anxiety.

The treatment of choice for social anxiety is cognitive behavioral therapy (CBT). Treatment is conducted both individually and in group-settings. Exposure therapy is central to CBT and is very effective in fear reduction.

In vivo exposure is effective when treating SAD, but conducting in vivo exposure in session can be challenging because relevant social situations might be difficult to obtain and control. In addition, finding the right setting for exposure can be time consuming and costly.

Exposure in virtual reality has several advantages compared to in vivo exposure. Virtual reality provides readily available environments for exposure, such as a meeting room with a group of people waiting for the patient to give a presentation. Furthermore, exposure in VR is highly controllable and can be modified to fit the needs of the patient. Finally, exposure takes place in confidentiality within the safety of the therapy room and thus the threshold for initiating exposure might be lower than for in vivo exposure.

AIMS AND HYPOTHESES

Primary hypothesis:

At post treatment the investigators expect that CBT including exposure therapy using individually tailored VR-content and a system to track anxiety levels (CBT-ExpVR) will result in lower levels of social anxiety than CBT with exposure in vivo (CBT-Exp). The outcome on social anxiety will be measured using the total score on Social Interaction Anxiety Scale (SIAS).

Secondary hypotheses:

At 6 and 12 months follow-up, the investigators expect that VR-treatment will result in lower levels of social anxiety than in vivo-treatment.

Post treatment and at 6 and 12 months follow up the investigators expect that VR-treatment will result in lower levels of depression and higher levels of self-rated health than in vivo-treatment.

The dropout rate the investigators expect will be lower for the VR-treatment compared to the in vivo-treatment.

In addition to the evaluation of effect, a health economic evaluation will be made from a societal perspective.

METHODS

Design:

The trial is a randomized controlled, assessor-blinded, parallel-group superiority trail. The study is conducted at Centre for Telepsychiatry in the Mental Health Services in the Region of Southern Denmark

Participants and recruitment:

Participants are referred to the trial's website where they are provided with written information about the study and are invited to complete online questionnaires screening for social anxiety symptoms and symptoms of depression. The questionnaire consists of Social Interaction Anxiety Scale and Major Depression Inventory and questions on current treatment and use of medication. Cut-off score for inclusion is <22 on SIAS and cut-off score for exclusion on MDI is >29. The online questionnaire might be supplemented by a phone call to inquire further information on current treatment and medication. No information will be obtained from patient records.

Eligible participants are invited to an assessment at Centre for Telepsychiatry. The assessment will be carried out using the short version of the Present State Examination. Participants who meet the inclusion criteria will be offered to participate in the study. Before the pre-treatment assessment, included patients will be asked to complete an informed consent form.

Randomization:

Participants are block randomized (1:1) using random block size. The block sizes will not be disclosed, to ensure concealment. Computer generated random numbers using the platform Sealed Envelope (www.sealedeenvelope.com) will be used to generate the allocation sequence. The allocation sequence is handled by a data manager from the Patient data Explorative Network (OPEN) and is unavailable to those who enroll and assign participants.

Blinding:

Psychologist responsible for the diagnostic interview are blind to treatment assignment. Participants are blinded to their treatment assignment until their first treatment session. Participants will only be blind to treatment assignment at the pre-test but not at later assessments. A clinician blind to treatment assignment will administer the assessment taking place at pre-test, mid-test, and post-test.

Sample size:

A recent study reported approximately 10-point drop in SIAS for standard treatment involving CBT and 20-point drop for CBT with virtual exposure with standard deviations around 15 points. A drop of 13 points on SIAS is considered reliable change.

If 35 participants are recruited for each group, this will lead to a statistical power of 0.80 comparing the VR-treatment to in vivo-treatment at the 0.05 significance level. To consider a 20% dropout the investigators plan to invite 90 participants in total.

Fidelity:

The interventions are manualized to increase treatment fidelity. To ensure that the treatment is delivered consistently and reliably in accordance with the manual the therapist will after each treatment session answer a self-report questionnaire on specific treatment targets for each session.

Data collection and management:

Data collected from the participants using self-report measures and data reported by therapist are collected using REDCap (Research Electronic Data Capture). To ensure confidentiality assigned researchers and the data manager at OPEN will be the only people with access to data at REDCap. Informed consent forms will be scanned and stored in REDCap . Data is stored at OPEN's server located in the Regions of Southern Denmark. Subjective Units of Distress Scale, Heart Rate, Electrodermal activity, and estimated anxiety are collected using iMotions, and data is saved on a secure folder on SharePoint.

Statistical analyses:

The primary statistical analysis will be carried out as intention to treat (ITT). The investigators will use linear mixed models to analyze the data. Separate analysis will be performed for each outcome variable. The investigators will use a two-level model with observations nested within participants. The fixed effects will be time, intervention, and the interaction between time and intervention as well as the baseline score. In addition to the primary analysis, a per-protocol analysis will be carried out on those participants completing at least 50% of the exposure sessions.

A sensitivity analysis will be carried out where missing data will be handled by multiple imputation (m=100). Imputations will be based on baseline characteristics and secondary outcome measures using chained equations. The moderating effect of the working alliance, depressive symptoms, alcohol and drug use on the treatment outcome will be explored as subgroup analysis with continuous moderators by including them as covariates interacting with treatment and time.

Model validation in the linear mixed model will be performed by inspection of QQ-plots of residuals and BLUPs (best linear unbiased predictors) to assess normality, and plotting residuals against fitted values to check homoscedasticity. If assumptions are violated, analysis will be performed after log-transformation. If assumptions do not hold on log-scale, bootstrapping will be applied.

Monitoring:

Cybersickness similar to motion sickness may occur in the VR-setting. Cybersickness will be monitored using the Simulator Sickness Questionnaire. Adverse events will be registered by the therapists.

Dissemination policy:

Results will be disseminated regardless of the magnitude or direction of effect. Both positive, negative, and inconclusive results will be made public and both beneficial and harmful effects of adaptive virtual reality exposure therapy will be reported. Dissemination will happen in scientific journals, at scientific conferences, as well as via www.clinicaltrials.gov. Authorship will be determined according to the Vancouver Guidelines

ELIGIBILITY:
Inclusion Criteria:

* Sufficient knowledge of the Danish Language.
* Fulfilling the diagnostic criteria for SAD according to ICD-10 classification of mental and behavioral disorders (F 40.1).

Exclusion Criteria:

* Previously diagnosed with autism spectrum disorders.
* Previously diagnosed with psychotic disorders.
* Severe depression (>29 Major Depression Inventory)
* Dependence syndrome
* Suicidal ideation.
* Dementia/Intellectual disability.
* Epilepsy.
* Taking part in other kinds of psychological intervention for SAD.
* Medication (SSRI, benzodiazepine, MAOI) type and doses needs to be stable three months prior to inclusions and during the intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
Social Anxiety Interaction Scale | post-treatment (week 10)
  The instrument is a measure of social anxiety symptoms and consists of 20 items assessing cognitive, affective, and behavioral responses to social interaction. The scale ranges from 0 to 80. Higher scores indicate worse outcome. Participants have to indicate to what degree they feel each statement is characteristic to them using a 5-point Likert scale (0 = not at all, 1 = slightly, 2 = moderately, 3 = very, 4 = extremely). The instrument has high internal consistency, Cronbach's alpha = 0.93, and high test-retest reliability, r = 0.92 (45).

SECONDARY OUTCOMES:
Leibowitz Anxiety Scale - Self report version | post-treatment (week 10)
  Leibowitz Anxiety Scale - Self report version is a measure of anxiety and avoidance in a range of social situations.
Fear of Negative Evaluation - Brief version | post-treatment (week 10)
  Fear of Negative Evaluation - Brief version is a measure of distress experiences when getting negative evaluations by others.
Major Depression inventory | post-treatment (week 10)
  Major Depression inventory is a measure of symptoms severity in depression.
EQ-5D-5L | post-treatment (week 10)
  EQ-5D-5L is a measure of health status.
Alcohol Use Disorders Identification Test | pre-treatment (week 1)
  Alcohol Use Disorders Identification Test is a screening for unhealthy alcohol use.
Drug use disorders identification test | pre-treatment (week 1)
  Drug use disorders identification test is a screening instrument for drug-related problems.

CONTACTS AND LOCATIONS:
Overall Officials: Per Trads Ørskov, Ph.d., Principal Investigator — Region of Southern Denmark
Locations (1):
- Centre for Telepsychiatry, Odense C, Denmark/Region of Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be stored on a server located in the Region of Southern Denmark. February 2025 data will be transferred to The Danish National Archives. Data are available upon reasonable request. Restrictions apply to the availability of data and approval is needed from Danish Data Protection Agency and or The Danish National Archives.
Supporting Information: Study Protocol
Time Frame: February 2025
Access Criteria: Restrictions apply to the availability of data and approval is needed from Danish Data Protection Agency and or The Danish National Archives.

REFERENCES:
- [Background] Organization, W. H. (1992). The ICD-10 classification of mental and behavioural disorders: clinical descriptions and diagnostic guidelines, World Health Organization.
- [Background] Ruscio AM, Brown TA, Chiu WT, Sareen J, Stein MB, Kessler RC. Social fears and social phobia in the USA: results from the National Comorbidity Survey Replication. Psychol Med. 2008 Jan;38(1):15-28. doi: 10.1017/S0033291707001699. Epub 2007 Nov 2. PMID 17976249
- [Background] Crome E, Grove R, Baillie AJ, Sunderland M, Teesson M, Slade T. DSM-IV and DSM-5 social anxiety disorder in the Australian community. Aust N Z J Psychiatry. 2015 Mar;49(3):227-35. doi: 10.1177/0004867414546699. Epub 2014 Aug 13. PMID 25122449
- [Background] Stein MB, Roy-Byrne PP, Craske MG, Bystritsky A, Sullivan G, Pyne JM, Katon W, Sherbourne CD. Functional impact and health utility of anxiety disorders in primary care outpatients. Med Care. 2005 Dec;43(12):1164-70. doi: 10.1097/01.mlr.0000185750.18119.fd. PMID 16299426
- [Background] Beesdo K, Bittner A, Pine DS, Stein MB, Hofler M, Lieb R, Wittchen HU. Incidence of social anxiety disorder and the consistent risk for secondary depression in the first three decades of life. Arch Gen Psychiatry. 2007 Aug;64(8):903-12. doi: 10.1001/archpsyc.64.8.903. PMID 17679635
- [Background] Heimberg RG, Stein MB, Hiripi E, Kessler RC. Trends in the prevalence of social phobia in the United States: a synthetic cohort analysis of changes over four decades. Eur Psychiatry. 2000 Feb;15(1):29-37. doi: 10.1016/s0924-9338(00)00213-3. PMID 10713800
- [Background] Bouchard S, Dumoulin S, Robillard G, Guitard T, Klinger E, Forget H, Loranger C, Roucaut FX. Virtual reality compared with in vivo exposure in the treatment of social anxiety disorder: a three-arm randomised controlled trial. Br J Psychiatry. 2017 Apr;210(4):276-283. doi: 10.1192/bjp.bp.116.184234. Epub 2016 Dec 15. PMID 27979818
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Olsen LR, Jensen DV, Noerholm V, Martiny K, Bech P. The internal and external validity of the Major Depression Inventory in measuring severity of depressive states. Psychol Med. 2003 Feb;33(2):351-6. doi: 10.1017/s0033291702006724. PMID 12622314
- [Background] Mattick RP, Clarke JC. Development and validation of measures of social phobia scrutiny fear and social interaction anxiety. Behav Res Ther. 1998 Apr;36(4):455-70. doi: 10.1016/s0005-7967(97)10031-6. PMID 9670605
- [Background] Tavoli A, Melyani M, Bakhtiari M, Ghaedi GH, Montazeri A. The Brief Fear of Negative Evaluation Scale (BFNE): translation and validation study of the Iranian version. BMC Psychiatry. 2009 Jul 9;9:42. doi: 10.1186/1471-244X-9-42. PMID 19589161
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Hildebrand M. The Psychometric Properties of the Drug Use Disorders Identification Test (DUDIT): A Review of Recent Research. J Subst Abuse Treat. 2015 Jun;53:52-9. doi: 10.1016/j.jsat.2015.01.008. Epub 2015 Jan 31. PMID 25682718
- [Background] Kennedy, R. S., Lane, N. E., Berbaum, K. S., & Lilienthal, M. G. (1993). Simulator Sickness Questionnaire: An enhanced method for quantifying simulator sickness. The International Journal of Aviation Psychology, 3(3), 203-220. https://doi.org/10.1207/s15327108ijap0303_3
- [Background] Horvath, A. O., & Greenberg, L. S. (1989). Development and validation of the Working Alliance Inventory. Journal of Counseling Psychology, 36(2), 223-233. https://doi.org/10.1037/0022-0167.36.2.223
- [Background] Robillard G, Bouchard S, Dumoulin S, Guitard T. The development of the SWEAT questionnaire: a scale measuring costs and efforts inherent to conducting exposure sessions. Stud Health Technol Inform. 2011;167:105-10. PMID 21685650
- [Derived] Orskov PT, Lichtenstein MB, Ernst MT, Fasterholdt I, Matthiesen AF, Scirea M, Bouchard S, Andersen TE. Cognitive behavioral therapy with adaptive virtual reality exposure vs. cognitive behavioral therapy with in vivo exposure in the treatment of social anxiety disorder: A study protocol for a randomized controlled trial. Front Psychiatry. 2022 Oct 10;13:991755. doi: 10.3389/fpsyt.2022.991755. eCollection 2022. PMID 36299540